CLINICAL TRIAL: NCT05964491
Title: Video Resources for People With Chronic Obstructive Pulmonary Disease: An Exploratory Qualitative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teesside University (Other)
Collaborators: International Primary Care Respiratory Group (Unknown)
Responsible Party: Principal Investigator, Kirsti Loughran, Research Fellow, Teesside University
Other Study IDs: 10857
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention studied

SUMMARY:
The IPCRG & Teesside University have searched the internet for video self management content for people living with COPD. Resources were reviewed by healthcare professionals and developed into a digital magazine to support people living with chronic obstructive Pulmonary Disease (COPD). The aims of this study are to

1. evaluate the use of the digital magazine format with video self-management content from an end user perspective, including

   1. what characteristics a good video resource should have
   2. what information is important to people with COPD to include in videos and digital magazines,
   3. the useability of a digital magazine format
2. Explore the opinions, experiences and preferences of people living with COPD for accessing online self-management content including barriers and facilitators for accessing online self-management video content

DETAILED DESCRIPTION:
The use of online sources of information for chronic disease management has steadily increased over recent years as technology becomes more intertwined with healthcare 1-3. Older adults, including those with COPD are now more likely to access online based video resources for information and advice on how to help their symptoms and health related quality of life using smart phones and tablets 2. During the Covid-19 pandemic many healthcare services, patient support groups and individuals living with chronic diseases produced video content that is freely accessible online 4. A recent project by the IPCRG to curate evidence-based video resources into a digital magazine discovered that content quality varied vastly and gaps in resources still remained 5. With the growing use of online video resources there is a need to establish what video resources need to have in terms of content, quality and personal appeal for people living with COPD to successfully use at aid self-management 6,7. The digital magazine was created with the understanding that it would be accessible to those who were not digitally excluded and appeal to those who had adequate digital literacy skills, however there are people with COPD who are digitally excluded and have varying degrees of digital literacy skills 8,9. The magazine format was chosen to provide a recognisable and easily navigated format however, it is not clear what formats, access and literacy levels are necessary to support the use of online video resources, in particular this digital magazine-based collation of videos 8.

The aims of this study are to

1. evaluate the use of the digital magazine format with video self-management content from an end user perspective, including

   1. what characteristics a good video resource should have
   2. what information is important to people with COPD to include in videos and digital magazines,
   3. the useability of a digital magazine format
2. Explore the opinions, experiences and preferences of people living with COPD for accessing online self-management content including barriers and facilitators for accessing online self-management video content

3-4 focus groups of ideally 4-8 people with COPD in each group will be conducted to discuss the use and make up of online self-management video content and wider experience of using online video resources for health information.

People with COPD will be recruited using the networks of those involved in the IPCRG project such as UK based support and exercise groups for people with COPD

Once returned, participants will be booked into online or face to face focus groups of around 4-8 people. Prior to attending to the focus groups, participants will be (1) asked to complete an eHEALS measure of digital literacy either over the phone with a researcher or return an electronic copy and (2) they will be requested to review a digital magazine.

The focus group will be facilitated by a researcher with experience in respiratory rehabilitation who has not been involved in developing the digital magazine based on a topic guide developed using extant literature and steering group discussions.

Focus groups would be transcribed verbatim and analysed by a steering group member with experience in respiratory rehabilitation and the researcher who facilitated the focus groups separately using NVivo software and an inductive thematic analysis approach 10. Themes will be discussed with a further researcher and finalised by consensus

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be anyone with a reported medical diagnosis of COPD, who is able to converse in English and has used a device to access the internet. Or the carers, partners or loved ones of someone living with COPD.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with a medically confirmed diagnosis of COPD or their carers, partners or loved ones.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative data | baseline
  Focus group transcripts

SECONDARY OUTCOMES:
eHEALS questionnaire | baseline
  Questionnaire about confidence finding and using electronic based health information

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No